CLINICAL TRIAL: NCT04126577
Title: Clinical Relevance of the Reverse Lipopolysaccharide Transport Pathway in Patients With Acute Peritonitis An Observational Prospective Study
Brief Title: Clinical Relevance of the Reverse Lipopolysaccharide Transport Pathway in Patients With Acute Peritonitis
Acronym: LIPS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: NGUYEN 2019
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Peritonitis
MeSH Terms: conditions — Peritonitis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with suspected peritonitis: Secondary peritonitis, sepsis and endotoxemia
  Interventions: Biological: blood samples

INTERVENTIONS:
Biological: blood samples — 4 blood samples of 6 ml each: one before the surgical incision, one after the operation, one 4h after the operation and the last 24h after the operation.

SUMMARY:
When there is infection in the intra-abdominal area, bacteria secrete toxins that are absorbed by the peritoneum. These toxins then bind to lipoproteins (which carry cholesterol in the blood) and are eliminated by the liver. Phospholipid transfer protein (PLTP) is a protein that facilitates the binding of bacterial toxins to lipoproteins and thus their elimination.

The objective of this study is to study the relationship between PLTP and the elimination of bacterial toxins in humans. A better understanding of the elimination of these toxins will lead to a better understanding of the disease. The ultimate objective is to improve the management of intra-abdominal infections.

ELIGIBILITY:
Inclusion Criteria:

* person who has given oral consent (patient or family member)
* pre-operative SEPSIS criteria (qSOFA >=2) or vasopressor or mechanical ventilation treatment
* admitted to the operating room for suspected generalized secondary peritonitis

Exclusion Criteria:

* person not affiliated to national health insurance
* person under legal protection (curatorship, guardianship)
* person under court order
* pregnant, parturient or breastfeeding woman
* minor
* immunosuppression (HIV infection, corticosteroid treatment > 0.15 mg/kg/day prednisolone equivalent > 2 weeks, immunosuppressive treatment, primary cellular immune deficiency)
* decision to limit or stop therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with secondary peritonitis, sepsis and endotoxemia
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
Perioperative plasma concentration in 3HM | 24 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France

REFERENCES:
- [Derived] Nguyen M, Alvarez M, Berthoud V, Pallot G, Abagri S, Leleu D, Pais-De-Barros JP, Ortega-Deballon P, Guinot PG, Masson D, Gautier T, Bouhemad B. High-density lipoproteins alleviate the endotoxin burden in patients with peritonitis and sepsis: The LIPS study. Eur J Clin Invest. 2025 Dec;55(12):e70099. doi: 10.1111/eci.70099. Epub 2025 Jul 19. PMID 40682387